CLINICAL TRIAL: NCT05301699
Title: Development and Validation of a Web-based Nomorgam to Predict Postoperative Complications After Radical Gastrectomy Among Elderly Gastric Cancer Patients
Brief Title: Development and Validation of a Web-based Nomorgam to Predict Postoperative Complications
Status: Completed | Type: Observational
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Xueyi Miao, Principal Investigator, Nanjing Medical University
Other Study IDs: XMiao
Record Dates: First submitted 2022-03-19; First posted 2022-03-31 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Gastric Cancer
Keywords: gastric cancer;postoperative complications;nomogram
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- training cohort: The training cohort was used for data analysis.
  Interventions: Other: data analysis; validating the nomogram
- validation cohort: The validation cohort was used for validating the nomogram
  Interventions: Other: data analysis; validating the nomogram

INTERVENTIONS:
Other: data analysis; validating the nomogram — Not Applicable. Our study did not involve intervention

SUMMARY:
The incidence of complications after gastrectomy remains high among elderly patients with gastric cancer. The investigators sought to establish and validate a web-based nomorgam for predicting total complications among elderly patients undergoing resection of gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with gastric cancer by endoscopy or pathology
* planned to receive radical surgery for the first time
* aged 60 or older

Exclusion Criteria:

* received preoperative radiotherapy or chemotherapy
* with other sites of malignant tumors

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: elderly gastric cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 582 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
postoperative complications during hospitalization | about 3 weeks
  the investigators captured it from electronic medical records

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing medical university, Nanjing, China

IPD SHARING:
Plan to Share IPD: Undecided